CLINICAL TRIAL: NCT04106128
Title: Prevalence, Impact and Reversibility of Acute Diaprhagmatic Dysfunction in Acute Respiratory Detresse Measured by Diaphragmatic Echogaphy
Brief Title: Prevalence, Impact and Reversibility of Acute Diaprhagmatic Dysfunction in Acute Respiratory Detresse
Acronym: PIRD-DRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-PP-15
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Distress Syndrome,Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound examination (Experimental): Assess the prevalence of acute diaphragmatic dysfunction by ultrasound
  Interventions: Diagnostic Test: ultrasound examination

INTERVENTIONS:
Diagnostic Test: ultrasound examination — Measuring the thickening fraction by diaphragmatic ultrasound of acute diaphragmatic dysfunction in patients admitted for acute respiratory distress

SUMMARY:
The diaphragm is a fine striated muscle with both extra respiratory and respiratory functions. It does most of the breathing work in interaction with the accessory respiratory muscles, the rib cage and the abdomen. Its activity can be measured by the transdiaphragmatic pressure generated by the magnetic stimulation of phrenic nerves (gold standard). It has been shown in the literature that diaphragmatic ultrasound, via the measurement of diaphragmatic excursion and especially the thickening fraction, is an easily accessible, non-invasive, reproducible and relevant technique for evaluating acute diaphragmatic dysfunction in resuscitation patients.

The objective of this project is to evaluate the prevalence of diaphragmatic dysfunction at admission in patients hospitalized in intensive care / respiratory intensive care unit for hypercapnic and/or hypoxic acute respiratory distress and requiring ventilatory support by non-invasive ventilation or high flow oxygen therapy. A subgroup analysis will then be carried out on 3 populations:

* Hypercapnic exacerbation of chronic obstructive pulmonary disease
* Hypoxic acute respiratory distress on infectious lung disease
* Acute pulmonary edema

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for acute respiratory distress management
* Etiological diagnosis either:
* Exacerbation of chronic obstructive pulmonary disease
* Infectious pneumonitis
* Acute pulmonary edema
* Need for a ventilatory support by either:
* Non-invasive ventilation
* High flow oxygen therapy (flow rate > 40L/min and oxygen inspired fraction > 40%)
* Mask oxygen therapy with flow rate > 5L/min

Exclusion Criteria:

* Exacerbation of interstitial pathology / pulmonary fibrosis
* Deformation of the thoracic cage
* Neurodegenerative pathology
* Need for oro-tracheal intubation from the beginning for mechanical ventilation
* Contraindication to Non-invasive Ventilation
* Patients undergoing diaphragmatic rehabilitation
* Immunocompromised patients
* History of known diaphragmatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Thickening fraction | 48 hours
  Measurement of the thickening fraction by diaphragmatic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Céline SANFIORENZO, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France